CLINICAL TRIAL: NCT04611087
Title: Self-Monitoring Focus Groups With Vibrant Lives Pasadena Participants
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA18-0407; NCI-2020-07542 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA18-0407 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Obesity-Related Malignant Neoplasm
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (focus group, interview): PHASE I: Participants attend 4 sessions of focus groups.
  PHASE II: Participants attend virtual Zoom interviews or one-on-one interviews.
  Interventions: Behavioral: Discussion; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Behavioral: Discussion — Attend focus groups
  Other Names: Discuss
Other: Interview — Attend interviews
Other: Survey Administration — Ancillary studies

SUMMARY:
This study investigates how individuals feel about a dietary mobile application. Information collected from focus groups and interviews may help doctors and mobile application developers to determine preferences and participant feedback about the appeal and usefulness of a mobile application.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To gather qualitative data to assess appeal, preference, and usefulness of a food and beverage self-monitoring mobile application.

OUTLINE:

PHASE I: Participants attend 4 sessions of focus groups.

PHASE II: Participants attend virtual Zoom interviews or one-on-one interviews.

ELIGIBILITY:
Inclusion Criteria:

* Pasadena Independent School District (ISD) employees who have completed the 6-month Vibrant Lives weight loss program or adults who have completed a weight loss program within the last 12 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have completed a weight loss program
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2018-07-03 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Preferences of food and beverage self-monitoring methodology and respective feedback messages | Up to 3 years
  Thematic and narrative analyses will be conducted from the transcriptions to gain an understanding for the preferences of food and beverage self-monitoring methodology and respective feedback messages.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Basen-Engquist, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org